CLINICAL TRIAL: NCT06399224
Title: Effect of Planter Vibration and Otago Exercise on Risk of Fall and Quality of Life in Hemiplegic Elderly
Brief Title: Effect of Planter Vibration and Otago Exercise in Old Hemiplegic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sandra Aziz Guirguis, Doctor of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vibration on hemiplegia
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Balance Disorders
Keywords: Hemiplegic elderly

STUDY DESIGN:
Intervention Model Description: The study group will be treated with both plantar vibration and Otago exercise whereas the control group will receive Otago exercise only. Both groups will receive a 50 minutes of otago exercise program except for the study group will take 15 minutes of plantar vibration with frequency of 80 Hz, with 10 seconds of vibration and 5 seconds of rest with total time 15 min before the Otago exercise. The frequency of the exercise will be 3 times a week for 12 weeks.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Planter vibrator with otago exercise (Active Comparator): This group will receive15 minutes of plantar vibration with frequency of 80 Hz, with 10 seconds of vibration and 5 seconds of rest with total time 15 min before the 50 minutes Otago exercise. The frequency of the exercise will be 3 times a week for 12 weeks.
  Interventions: Device: Local Plantar vibrator; Other: Otago exercise
- Otago exercise (Active Comparator): This group will receive 50 minutes Otago exercise only. The frequency of the exercise will be 3 times a week for 12 weeks.
  Interventions: Other: Otago exercise

INTERVENTIONS:
Device: Local Plantar vibrator — A vibrating device that applies 80 hz vibration waves applied on the sole of the foot
  Other Names: Vibrasens (Techno Concept, Loupian, France)
  Arms: Planter vibrator with otago exercise
Other: Otago exercise — Warm up Front Knee strength Back knee strength Side hip strength Calf raising Toe raising Sit to stand Heel walk Toe walk One leg standing Side way walk Cool down

SUMMARY:
This study aims to determine effect of Plantar vibration and Otago exercise on risk of fall and quality of life in hemiplegic elderly

DETAILED DESCRIPTION:
Stroke is one of the major causes of permanent disability. Stroke can have many causes and occurs mainly in old age, Hemiplegic patients have a two-fold higher risk of falling than other patients of the same age or gender, beside fall in older adults can cause significant physical and psychological injury to the individual. Otago exercises are the interventions given for fall prevention in elderly and showed good results with hemiplegic cases as well, it is easy and could be done by old adults even at home. Plantar vibration as a cheap, portable, and easy applicable, saving time and with no effort could be a good choice as a treatment tool to be added for old hemiplegic patients treatment programme. Thus applying an easy and effective programme for old hemiplegic subjects that reduces their risk of fall and improves their balance and ADL and at the same time helps them to conduct it easily and adhere to it should be our target to full fill.

ELIGIBILITY:
Inclusion Criteria:

* first-ever stroke
* age 65-75years
* duration since stroke ≥6 months
* balance deficit confirmed by one leg stance (OLS) test; patient unable to stand on affected leg for 30s with eyes open
* able to walk without the use of aids .able to understand verbal commands.

Exclusion Criteria:

* participation in other treatment protocols for balance
* presence of conditions other than stroke affecting balance
* history of lower-limb surgery within the previous year
* fixed ankle contractures
* cognitive impairments (MMSE<24)

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | Through 12 weeks
  It is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete.
Time up and go test | Through 12 weeks
  The participant was instructed to sit back in the chair without arms, to stand up on the command "Go," walk 3 m to the line marked on the floor at a normal pace, turn 180°, and walk back to the chair, and sit down again on the chair,An older adult who takes ≥12 seconds to complete the TUG is at risk for falling.

SECONDARY OUTCOMES:
Stroke specific quality of life scale | Through 12 weeks
  It is a patient-centered outcome measure intended to provide an assessment of health-related quality of life (HRQOL) specific to patients with stroke.Patients must respond to each question of the SS-QOL with reference to the past week. It is a self-report scale containing 49 items in 12 domains.Higher scores indicate better functioning.
Modified barthel index | Though 12 weeks
  It is composed of the following 10 items investigating 10 functional ADLs: feeding, personal hygiene, bathing, dressing, chair-bed transfer, toileting, bladder continence, bowel continence, ambulation or wheelchair use, and stair climbing. The score for each item is attributed by the clinician who observes the patient while performing the functional task and evaluates the amount of assistance the patient requires using a 5-point Likert scale.Each activity is assigned a score from 0 to 15, indicating the patient's level of independence.Higher scores signify greater independence, while lower scores indicate dependence or the need for assistance.
Ankle PROM | Though 12 weeks
  The 90° was defined as the neutral position for the measurements using an ankle biplane goniometer Ankle dorsiflexion and plantarflexion from the neutral position was given either a positive or negative value

CONTACTS AND LOCATIONS:
Overall Officials: A.M Baky, Professor, Study Director — faculty of physical therapy
Locations (1):
- Faculty of physical therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khalifeloo M, Naghdi S, Ansari NN, Akbari M, Jalaie S, Jannat D, Hasson S. A study on the immediate effects of plantar vibration on balance dysfunction in patients with stroke. J Exerc Rehabil. 2018 Apr 26;14(2):259-266. doi: 10.12965/jer.1836044.022. eCollection 2018 Apr. PMID 29740561
- [Background] Yang Y, Wang K, Liu H, Qu J, Wang Y, Chen P, Zhang T, Luo J. The impact of Otago exercise programme on the prevention of falls in older adult: A systematic review. Front Public Health. 2022 Oct 20;10:953593. doi: 10.3389/fpubh.2022.953593. eCollection 2022. PMID 36339194